CLINICAL TRIAL: NCT00457795
Title: 24-hour IOP-lowering Effect of Brimonidine 0.1%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-080806-2
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-10

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Brimonidine Tartrate

ARMS (1):
- brimonidine 0.1% (Experimental): brimonidine 0.1%
  Interventions: Drug: brimonidine 0.1% (Alphagan® P)

INTERVENTIONS:
Drug: brimonidine 0.1% (Alphagan® P) — Brimonidine 0.1%, 1 drop three-times daily for 4 weeks
  Other Names: Alphagan® P

SUMMARY:
This study will evaluate the efficacy and safety of brimonidine 0.1% three-times daily in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* patients with open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* allergy to brimonidine
* inability to complete 24 hour stay for monitoring

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Allergan
Locations (1):
- San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brimonidine 0.1%
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Brimonidine 0.1%
Number analyzed (Participants) | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 58.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) for a 24-Hour Period at Week 4
Description: IOP for a 24-hour period separated into diurnal(7AM-11PM or awake period) and nocturnal (11PM-7AM or sleep period) at week 4. IOP is a measurement of the fluid pressure inside the eye. Measurements of IOP were taken in the sitting and supine (laying down face up) body positions during the 16-hour diurnal (awake) period and in the supine position during the 8-hour nocturnal (sleep) period.
Time Frame: Week 4
Population: Intent to Treat defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Brimonidine 0.1%
Number analyzed (Participants) | 15
Millimeters of mercury (mmHg)
  Diurnal IOP Sitting at Week 4 | 16.8 (2.8)
  Diurnal IOP Supine at Week 4 | 21.1 (2.3)
  Nocturnal IOP Supine at Week 4 | 23.0 (2.8)

2. Secondary Outcome: Change From Baseline in Intraocular Pressure (IOP) for a 24-Hour Period at Week 4
Description: Change from baseline in IOP for a 24-hour period separated into diurnal (7AM-11PM or awake period) and nocturnal (11PM-7AM or sleep period) at week 4. IOP is a measurement of the fluid pressure inside the eey. Measurements of IOP were taken in the sitting and supine (laying down face up) body positions during the 16-hour diurnal (awake) period and in the supine position during the 8-hour nocturnal (sleep) period. A negative number change from baseline indicates an improvement.
Time Frame: Baseline, Week 4
Population: Intent to Treat defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Brimonidine 0.1%
Number analyzed (Participants) | 15
Millimeters of mercury (mmHg)
  Diurnal IOP Sitting at Baseline | 19.2 (2.7)
  Diurnal IOP Supine at Baseline | 23.1 (2.1)
  Nocturnal IOP Supine at Baseline | 22.7 (2.6)
  Diurnal IOP Sitting Change from Baseline at Week 4 | -2.4 (1.4)
  Diurnal IOP Supine Change from Baseline at Week 4 | -1.9 (1.3)
  Nocturnal IOP Supine Change from Baseline at Wk 4 | 0.3 (1.9)

3. Secondary Outcome: Ocular Perfusion Pressure (OPP) for a 24-Hour Period at Week 4
Description: Ocular perfusion pressure (OPP) calculated for a 24-hour period separated into diurnal (7AM-11PM or awake period) and nocturnal (11PM-7AM or sleep period) at week 4. Ocular perfusion pressure is blood pressure minus the intraocular pressure, which is a measurement of the fluid pressure inside the eye. Measurements of IOP and blood pressure were taken in the sitting and supine (laying down face up) body positions during the 16-hour diurnal (awake) period and in the supine position during the 8-hour nocturnal (sleep) period.
Time Frame: Week 4
Population: Intent to Treat defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Brimonidine 0.1%
Number analyzed (Participants) | 15
Millimeters of mercury (mmHg)
  Diurnal OPP Sitting at Week 4 | 46.8 (7.6)
  Diurnal OPP Supine at Week 4 | 53.8 (9.8)
  Nocturnal OPP Supine at Week 4 | 49.2 (11.2)

4. Secondary Outcome: Change in Ocular Perfusion Pressure (OPP) Over a 24-Hour Period at Week 4
Description: Change in ocular perfusion pressure (OPP) calculated over a 24-hour period separated into diurnal (7AM-11PM or awake period) and nocturnal (11PM-7AM or sleep period) at Week 4. Ocular perfusion pressure is blood pressure minus the intraocular pressure, which is a measurement of the fluid pressure inside the eye. Measurements of IOP and blood pressure were taken in the sitting and supine (laying down face up) body positions during the 16-hour (awake) period and in the supine position during the 8-hour nocturnal (sleep) period.
Time Frame: Week 4
Population: Intent to Treat defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Brimonidine 0.1%
Number analyzed (Participants) | 15
Millimeters of mercury (mmHg)
  Diurnal Change in OPP Sitting at Week 4 | 1.1 (5.6)
  Diurnal Change in OPP Supine at Week 4 | 0.3 (4.9)
  Nocturnal Change in OPP Supine at Week 4 | -3.0 (6.1)

ADVERSE EVENTS:
Arm/Group | Brimonidine 0.1%
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo